CLINICAL TRIAL: NCT06175078
Title: Investigation of Three-Dimensional Ultrasound Imaging and Spectroscopy for Characterizing Breast Masses
Brief Title: Three-Dimensional Ultrasound Imaging and Spectroscopy for Characterizing Breast Masses
Status: Not yet recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 5587
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Breast Masses
Keywords: Ultrasound Imaging 3D; Spectroscopy
MeSH Terms: conditions — Breast Neoplasms | interventions — Spectrum Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with suspected breast cancer: Patients with suspected breast cancer will be recruited and scanned for this study. The results of ultrasound data analysis will be compared and correlated to the histopathology reports on routine core biopsy specimens, surgery reports, or radiology reports.
  Interventions: Device: Ultrasound Imaging 3D and Spectroscopy

INTERVENTIONS:
Device: Ultrasound Imaging 3D and Spectroscopy — Ultrasound imaging and spectroscopy will consist of collecting three dimensional data. Regions of interest in each of the tumour images and in the adjacent normal tissue will be selected for analysis.

SUMMARY:
The purpose of the study is to test the hypothesis that quantitative ultrasound techniques including spectroscopy may be used as a non-invasive biomarker for characterization of suspected breast cancers. The main goal is to select and identify an optimal set of quantitative ultrasound parameters that can be used, non-invasively, to characterize suspected breast cancers, as identified based on the histopathology reports on core biopsy specimens, surgery reports, or radiology reports. Primary endpoint will correlate quantitative ultrasound parameters to the histopathological properties, as determined from pathology reports on core biopsy specimens, surgery reports, or radiology reports. The secondary endpoint in this study will include correlating the results of ultrasound-based breast cancer characterization with 2 and 5-years clinical outcomes.

DETAILED DESCRIPTION:
This project is an observational/early validation study in human subjects that will use ultrasound imaging and spectroscopy to characterize suspected breast cancers. Patients will be imaged with ultrasound, and the acquired data will be analyzed using quantitative ultrasound techniques, in conjunction with textural analysis on generated parametric images. Results of quantitative ultrasound data analysis for these breast lumps will be compared to and correlated with histopathological characteristics from pathology reports on core biopsy specimens, surgery reports, or radiology reports.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men with suspected breast cancer
2. Patients should have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks prior to registering in the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration.
2. Receiving any other investigational agents.
3. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women or men with suspected breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of quantitative ultrasound parameters to the histopathological properties of suspected breast cancer tissues. | Up to 2 years
  As a primary endpoint, correlate changes in ultrasound backscatter parameters obtained using spectroscopic techniques, in conjunction with textural analysis on generated parametric images, to the histopathological characteristics from pathology reports on core biopsy specimens, surgery reports, or radiology reports.

SECONDARY OUTCOMES:
Correlating the results of ultrasound-based breast cancer characterization to clinical outcomes. | Up to 5 years
  The secondary endpoint in this study will include correlating the results of ultrasound-based breast cancer characterization with 2 and 5-years clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No